CLINICAL TRIAL: NCT00473980
Title: Preoperative Treatment With NSAID in Colorectal Cancer Patients in Relationship to Tumor Host Reactions
Brief Title: Preoperative Non-steroidal Anti-inflammatory Drugs(NSAID) to Colorectal Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kl4501122
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer
Keywords: MHC; CTLs; Colon carcinoma; NSAID; Survival
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Indomethacin; Celecoxib; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental): Treatment with indomethacin or celecoxib
  Interventions: Drug: Indomethacin, celecoxib, esomeprazole
- SHAM (Sham Comparator): Sham treatment
  Interventions: Drug: Indomethacin, celecoxib, esomeprazole

INTERVENTIONS:
Drug: Indomethacin, celecoxib, esomeprazole

SUMMARY:
The study is designed to evaluate effects of NSAIDs on immune activity inside and close to tumor tissue in patients with colorectal cancer.

DETAILED DESCRIPTION:
Study and control patients are randomized to receive preoperative treatment with indomethacin or celecoxib compared to sham treatment.Tumor biopsies are taken at operation and used for analyses of tumor immunity and gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Colon carcinoma scheduled for curative operation

Exclusion Criteria:

* Diabetes, steroid medication, liver and kidney impairment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1998-12; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Immune reactivity | Acute evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Kent Lundholm, MD, prof, Principal Investigator — Göteborg University
Locations (1):
- Department of Surgery, Gothenburg, Sweden

REFERENCES:
- See also: Göteborg University — http://www.gu.se